CLINICAL TRIAL: NCT06635785
Title: Safety, Pharmacokinetics, and Efficacy of AI-081, a Bispecific Antibody for PD-1 And VEGF in Advanced Solid Tumors
Acronym: BiPAVE-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BiPAVE-001
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AI-081 (Experimental): AI-081 will be given by IV infusion in designated dose, q3w.
  Interventions: Drug: AI-081

INTERVENTIONS:
Drug: AI-081 — AI-081 is a humanized monoclonal antibody targeting PD-1 and VEGF.
  Other Names: Bispecific anti-PD-1/VEGF

SUMMARY:
BIPAVE-001 is a Phase 1-2 study for evaluating the safety, pharmacokinetics (PK), and efficacy of AI-081 in solid tumors.

DETAILED DESCRIPTION:
AI-081 is a bispecific antibody against PD-1 and VEGF. The study BiPAVE-001 is consisting of two integrated parts: Part A is the first-in-human dose escalation study to determine the recommended Phase 2 dose (RP2D) of AI-081 monotherapy, while Part B are dose optimization trials comparing the safety and clinical activities of AI-081 at RP2D and one dose level lower than RP2D (RP2D-1), either as monotherapy or in combination therapy with standard of care (SOC) in selected indications.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age on the day of signing informed consent.
* Male or female, female patient of childbearing potential must have negative pregnancy test.
* Patient must have a performance status of ≤ 1 on the ECOG Performance Scale.
* Patients must have a histological or cytological diagnosis of solid tumors and have metastatic disease or locally advanced disease.
* Measurable disease as determined by RECIST 1.1
* Patient must have adequate organ function as indicated by the following laboratory values
* Patient has voluntarily agreed to participate by giving written informed consent.
* Female patients enrolled in the study, if having childbearing potential (WOCBP) and sexually active, must agree to use adequate and effective birth control starting with the first dose of study drug through 90 days after the last dose of study therapy.
* Male patients, if sexually active, must agree to use adequate and effective methods of contraception starting with the first dose of study drug through 90 days after the last dose of study therapy.

Exclusion Criteria:

* Patients who have not recovered to NCI CTCAE grade ≤ 1 from an adverse event (AE) due to cancer therapeutics except the chemotherapy-associated peripheral neuropathy (motor or sensory) or alopecia. Patients with ongoing and adequately controlled endocrine immune-related AEs are considered stable and eligible for enrollment. The washout period for treatment regimen containing monoclonal antibodies is 28 days. Palliative radiotherapy for painful metastases or metastases in potentially sensitive locations (e.g., epidural space) ≥ 7 days prior to the first dose of study drug. Best supportive care, such as thyroxine, insulin, steroid replacement treatment, blood transfusion and therapy for non-cancer condition are allowed.
* Patients who are currently enrolled in any other clinical trial testing an investigational agent or device, or with concurrent anticancer treatment (except palliative bone-directed radiotherapy), immune therapy, or cytokine therapy or anticipated to require another antineoplastic therapy during the study.
* Patients who are on chronic systemic steroid therapy at doses higher than 10 mg/day prednisone or equivalent within 7 days before first treatment.
* Patients who have brain metastases or leptomeningeal metastases.
* Patient with a different cancer other than the one treated under this protocol, which requires systemic treatments within 24 months prior to C1D1.
* Patient has history of grade ≥3 allergic or hypersensitivity to IV infusion medications, or severe allergic reactions to food, pollen, oral medications, or atopic dermatitis or asthmatic episodes that required hospitalization.
* Within past 6 months with history of significant cardiovascular acute myocardial infarction, acute coronary syndrome, ischemic or hemorrhagic stroke, revascularization procedures, acute pulmonary embolism or any disorders resulted in LVEF < 40% at the time of screening or colitis, small bowel obstruction, hepatitis or pancreatitis adrenal insufficiency, or severe immunotherapy related AE (irAE≥ grade 3).
* Patients who have acute infections which require systemic treatments within 14 days prior to C1D1.
* Patients who, in the opinion of the treating Investigator, have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or make study participation not in the best interest of the patient, in the opinion of the treating Investigator. Investigators should discuss the case with the Sponsor and/or study leaders.
* Patients with known psychiatric or substance abuse disorders may interfere with cooperation with the requirements of the trial.
* Patients who are pregnant or breastfeeding or plan pregnancy or fathering the child during the study or within 6 months after the last dosing of study drug
* Patients with tumor surrounds important blood vessels or has obvious necrosis, cavitation, or invades surrounding important organs and blood vessels or otherwise with high risk of fatal hemorrhage
* Uncontrolled hypertension: systolic pressure ≥ 150 millimeters of mercury (mmHg) or diastolic pressure ≥ 90 mmHg on repeated measurements that cannot be managed by standard antihypertension medications ≤ 28 days before the first dose of study drug(s).
* Medical history of cardiovascular diseases, gastrointestinal perforation or gastrointestinal fistula within 6 months prior to the first dose.
* Patients with clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage.
* With a history of interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung diseases, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 21 Days
  Maximal tolerable dose (MTD), the study drug, AI-081
Dose Limiting Toxicity (DLT) | 21 Days
  The number of subjects who have Dose limiting toxicity (DLT) as defined by protocol DLT criteria during the first cycle of study drug, AI-081, administration.

SECONDARY OUTCOMES:
Cmax of AI-081 | 63 Days
  The highest Serum concentration of AI-081 after IV infusion at cycle 1 and cycle 3 from different timepoints (within 60 minutes before dosing, 60 minutes post-dose, 6 hours post-dose, 24 hours post dose, day 8, 15 and 21 post-dose) after drug administration.
The serum half-life of AI-081 | 63 Days
  To determine the drug concentration in serum samples that are taken in various timepoints (Cycle 1 and Cycle 3: within 60 minutes before dosing, 60 minutes post-dose, 6 hours post-dose, 24 hours post dose, day 8, 15 and 21 post-dose. Cycle 2 and Cycle 4-13: within 60 minutes before dosing and 60 minutes post-dose) during the treatment in order to calculate drug half life.

CONTACTS AND LOCATIONS:
Overall Officials: Kai He, MD, PhD, Principal Investigator — The Ohio State University James Cancer Center
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Highlands Oncology Group, Springdale, Arkansas
  - University of Florida UF Health Cancer Center, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Ocala Oncology Center PL DBA Florida Cancer Affiliates, Ocala, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Norton Cancer Center, Louisville, Kentucky
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - The Tisch Cancer Institute, Mount Sinai Medical Center, New York, New York
  - University of North Carolina at Chapel Hill Cancer Center, Chapel Hill, North Carolina
  - Novant Health Cancer Institute, Winston-Salem, North Carolina
  - The Ohio State University James Cancer Center, Columbus, Ohio
  - Prisma Health, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No